CLINICAL TRIAL: NCT05498545
Title: A Clinical Study to Evaluate the Safety, Tolerability, and Efficacy of Universal BCMA-targeted LUCAR-B68 Cells Product in Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: Universal BCMA-targeted LUCAR-B68 Cells in Patients With Relapsed/Refractory Multiple Myeloma
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Collaborators: Nanjing Legend Biotech Co. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BM2L202201
Record Dates: First submitted 2022-08-10; First posted 2022-08-12 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Relapsed/Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LUCAR-B68 cells product (Experimental): Each subject will receive LUCAR-B68 cells
  Interventions: Biological: LUCAR-B68 cells product

INTERVENTIONS:
Biological: LUCAR-B68 cells product — Before treatment with LUCAR-B68 cells, subjects will receive a conditioning regimen

SUMMARY:
A Clinical Study to Evaluate the Safety, Tolerability, and Efficacy of Universal BCMA-targeted LUCAR-B68 Cells Product in Patients With Relapsed/Refractory Multiple Myeloma

DETAILED DESCRIPTION:
This is a prospective, single-arm, open-label, dose-finding and dose-expansion study that evaluates the safety, tolerability, PK, and anti-tumor efficacy of LUCAR-B68 cell preparations in relapsed/refractory multiple myeloma subjects who received adequate standard therapy

ELIGIBILITY:
Inclusion Criteria:

1. The subject voluntarily participates in the clinical study; Fully understand and be Informed of the study and sign the Informed consent (Informed Consent Form, ICF); Willing to follow and able to complete all test procedures; Informed consent must be obtained before initiating any tests or procedures related to the study that are not part of the standard treatment of the subject's disease;
2. Subjects ≥ 18 years of age.
3. Eastern Cooperative Oncology Group performance status score of 0, 1, or 2;
4. Documented initial diagnosis of MM according to IMWG diagnostic criteria.
5. Presence of measurable disease at screening.
6. Received a PI and an IMiD (except thalidomide).
7. Received at least 3 prior lines of therapy for multiple myeloma, undergone at least 1 complete cycle of treatment for each line, unless progressive disease (PD) was documented by IMWG criteria as the best response to the regimen. Also, subjects refractory or intolerant to any PI and any IMiD in their previous treatment afterwards are eligible.
8. Expected survival ≥ 3 months.
9. Clinical laboratory values meet screening visit criteria
10. Fertile women must be negative using a highly sensitive serum pregnancy test (β human chorionic gonadotropin [β -HCG]) at screening time and before initial treatment with cyclophosphamide and fludarabine;

Exclusion Criteria:

1. No response to prior BCMA-targeted CAR-T therapy (except in subjects who relapsed after CR to prior CAR-T treatment);
2. Prior treatment with any antibody targeting BCMA;
3. Known active, or prior history of central nervous system (CNS) involvement, or clinical signs of membrane/spinal membrane involvement of multiple myeloma;
4. Serious underlying medical conditions
5. Positive of any hepatitis B surface antigen (HBsAg), hepatitis B virus deoxyribonucleic acid (HBV DNA), hepatitis C antibody (HCV-Ab), hepatitis C virus ribonucleic acid (HCV RNA), human immunodeficiency virus antibody (HIV-Ab) at the time of screening;
6. Male subjects who have a birth plan during the study period or within 1 year after the study treatment
7. Female subjects who are pregnant, breast-feeding, or plan to become pregnant during the study period or within 1 year after the study treatment
8. The investigator considered that the subjects were not suitable for any conditions of participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Incidence, severity, and type of treatment-emergent adverse events (TEAEs) | Minimum 2 years after LUCAR-B68 infusion (Day 1
  An adverse event refers to any untoward medical occurrence in a clinical investigation subject administered a pharmaceutical product (investigational or non-investigational), which does not necessarily have a causal relationship with the treatment
Dose-limiting toxicity (DLT) rate | Minimum 2 years after LUCAR-B68 infusion (Day 1)
  Dose-limiting toxicity (DLT) refers to a drug-related toxicity during treatment with the drug, the severity of which is clinically unacceptable, limiting the further escalation of drug dose
Recommended Phase 2 dose (RP2D) finding | 30 days after LUCAR-B68 infusion (Day 1)
  RP2D established through ATD+BOIN design
CAR positive NK cells in peripheral blood and bone marrow | Minimum 2 years after LUCAR-B68 infusion (Day 1)
  CAR positive NK cells in peripheral blood and bone marrow after LUCAR-B68 infusion
CAR transgene levels in peripheral blood | Minimum 2 years after LUCAR-B68 infusion (Day 1)
  CAR transgene levels in peripheral blood after LUCAR-B68 infusion

SECONDARY OUTCOMES:
Overall response rate (ORR) | Minimum 2 years after LUCAR-B68 infusion (Day 1)
  The ORR is defined as the percentage of participants who achieve partial response (PR) or better according to international myeloma working group (IMWG) criteria
Duration of Response (DOR) | Minimum 2 years after LUCAR-B68 infusion (Day 1)
  Duration of response (DOR) will be calculated among responders (with a PR or better response) from the date of initial documentation of a response (PR or better) to the date of first documented evidence of progressive disease, as defined in the IMWG criteria or death due to any cause, whichever occurs first
Time to Response (TTR) | Minimum 2 years after LUCAR-B68 infusion (Day 1)
  Time to response (TTR) is defined as the time between date of the initial infusion of LCAR-B38M CAR-T cells and the first efficacy evaluation that the participant has met all criteria for PR or better
Progress Free Survival (PFS) | 2 years after LUCAR-B68 infusion (Day 1)
  Progression Free Survival (PFS) is defined as the time from the date of first infusion of the LUCAR-B68 to the first documented disease progression (according to IMWG criteria) or death (due to any cause), whichever occurs first
Overall Survival (OS) | Minimum 2 years after LUCAR-B68 infusion (Day 1)
  Overall Survival (OS) is defined as the time from the date of first infusion of LUCAR-B68 to death of the subject
Incidence of anti- LUCAR-B68 antibody | Minimum 2 years after LUCAR-B68 infusion (Day 1)
  Venous blood samples will be collected to measure LUCAR-B68 positive cell concentrations and the transgenic level of LUCAR-B68, at the time points when anti- LUCAR-B68 antibody serum samples are evaluated

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No